CLINICAL TRIAL: NCT05594966
Title: Neuroimaging Combining Biomarkers for Identifying Long-term Cognitive Dysfunction and Delirium After Cardiac Surgery Early and Availably
Brief Title: Neuroimaging Combining Biomarkers for Identifying Long-term Cognitive Dysfunction and Delirium
Acronym: NeuroIDEA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Peiying Li, Professor, RenJi Hospital
Other Study IDs: NeuroIDEA
Record Dates: First submitted 2022-10-23; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium; Cerebral Small Vessel Diseases; Covert Postoperative Stroke
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Cerebral Small Vessel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 5 ml peripheral venous blood samples will be taken before and after the surgery. The blood samples will be preserved in ethylenediaminetetraacetic acid tubes and patient's information and serial number will be recorded on the tube. Samples are centrifuged for 10min at 2000x g and the supernatants will be transformed into Eppendorf tubes and stored at -80 °C. DNA will be extracted according to the protocol. The DNA samples will be stored at -80°C until further use. Before taking blood from patients, the purpose of using blood samples will be fully explained to them and informed consent will be obtained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebral Small Vessel Disease: In this group, patients are diagnosed with cerebral small vessel disease preoperatively using multimodal MRI.
  Interventions: Diagnostic Test: multimodal MRI
- non-Cerebral Small Vessel Disease: In this group, cerebral small vessel disease is ruled out by preoperative multimodal MRI.
  Interventions: Diagnostic Test: multimodal MRI

INTERVENTIONS:
Diagnostic Test: multimodal MRI — patients are diagnosed with cerebral small vessel disease preoperatively using multimodal MRI

SUMMARY:
Postoperative Cognitive Dysfunction(POCD) is commonly seen in cardiac surgery, which may lead to poor pognosis. Cerebral small vessel disease(CVSD) is refer as the main resource of delirium among elderly people. In the study, CVSD will be diagnosed using multimodal MRI. And we want to select a high correlating COPD biomarker through CyTOF. We also want to investigate a medical model to select the high risk patients who may suffer from POCD after cardiac surgery.

DETAILED DESCRIPTION:
This study will investigate whether preoperative CSVD and CyTOF will help to predict the occurencce of Postoprative Cognitive Dysfunction(POCD) in 1 year after surgery. The investigators perform a prospective cohort study among selective cardiac surgery patients between 50 to 85 years old. All participates have pre-operative head multimodel MRI in Renji Hospital Affiliated to Shanghai Jiaotong University. Incusion and exclusion criteria and relevant data were collected. Patients' age, gender, specific surgical methods, educational background, BMI, tobacco and alcohol history, and systematic medical history were collected before surgery, specific history (heart disease, heart failure, arrhythmia, cornoary artery stent implantation, and history of cardiac surgery), medical history (blood pressure medication, anti-arrhythmic drugs, diuresis, anti-arrhythemic drugs, diuresis, anticoagulant drugs), laboratory examination, auxiliary examination(blood routine, blood coagulation, liver and kidney function, etc.), and Cognitive Function Assessment Scale(MMSE, MOCA, ADL, GDSS). Perioperative indicators were also collected, including use of anesthetics, anestetic time,vital signs, etc. Blood sample should be taken before and after surgery. Postopeative data including: POD whithin 5 days after surgery, cardiovascular drugs use in ICU, mechanical ventilation time, length of stay in ICU, occurrence of complicatiosns of patients, Cognitive function Assessment Scale 1 year after surgery. POD was assessed by a professionally trained clinician twice daily at 8-12 hour intervals, using CAM-ICU scale, if diagnosis with POD, DRS-98 is used to evaluate th severity of POD. POCD was assessed by a professionally trained clinican at 1 year after surgery. The incidence of POD and POCD was analyzed between groups, and the association between each index and delirium and POCD was analyzed by logistic regresssion. The waste blood from routine peripheral blood examination was collected before operation, at the end of operation, on the second day after operation and one year after opertion for the detection of biomarkers by CyTOF, and the composite model of MRI and biomarkers was established.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 50 years to 85 years;
2. The patient is going to have selective cardiac surgery;
3. Written informed consent is obtained before the surgery.

Exclusion Criteria:

1. mental illness;
2. Already have other diseases that can cause dementia, such as Alzheimer's disease, Lewy body dementia, Frontotemporal dementia, progressive supranuclear palsy, Parkinson's disease, Creutzfeldt-Jakob disease, Huntington's disease, alcohol and drug dependence, Neurosyphilis, systemic lupus erythematosus; or preoperative MRI shows hippocampal and temporal lobe atrophy more than three levels
3. Have suffered from other brain diseases (such as overt stroke, multiple sclerosis, central nervous system infection with sequelae, etc.);
4. Preoperative MRI indicates covert stroke MMSE or MoCA scale cannot be completed due to other reasons (such as hearing impairment or visual impairment)
5. MRI contraindications before or after surgery or patients who cannot tolerate MRI imaging
6. Stage 3 or 4 malignant tumors, and high malignancy and poor prognosis cancer, such as pancreatic cancer, gallbladder cancer, and bile duct cancer.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The incidence of POCD after cardiac surgery varies greatly in different studies. Accroding to JAMA and Lancet papers, the incidence of POCD in patients one year after cardiac surgeries is 20-31%. According to the Events per Variable method, the main objective model establishment will explore 5 Events of independent variables. Assuming EPV is 10, the incidence of POCD is 26%, so the number of POCD patients after surgeries should be 5*10=50. Take 10% loss of follow-up rate into account, the total sample size required is 50/26%*110%=211
Sampling Method: Non-Probability Sample
Enrollment: 211 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
A medical model to predict the POCD after cardiac surgery. | 1 year
  A composite model of MRI and biomarker risk factors to predict the incidence of POCD in patients undergoing selective cardiac surgery

SECONDARY OUTCOMES:
Build a medical model to predict the POD after cardiac surgery. | 5 days
  A composite model of MRI and biomarker risk factors to predict the incidence of POD in patients undergoing selective cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Li Peiying, MD, Principal Investigator — chief professor of Anesthesiology Departmetn,Renji Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University, School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared starting 6 months after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All the IPD and any additional supporting information will become available starting 6 months after publication for at least 5 years.
Access Criteria: Requests to access all the IPD and additional supporting information will be addressed and reviewed by the corresponding author of the related publication. Access criteria include that the requests shall be submitted by a researcher on an institutional headed paper; the requests shall come with all the detailed contact information of the researcher and the administration office of the institution.

REFERENCES:
- [Result] Wardlaw JM, Smith C, Dichgans M. Small vessel disease: mechanisms and clinical implications. Lancet Neurol. 2019 Jul;18(7):684-696. doi: 10.1016/S1474-4422(19)30079-1. Epub 2019 May 13. PMID 31097385
- [Result] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200
- [Result] Guenther U, Theuerkauf N, Frommann I, Brimmers K, Malik R, Stori S, Scheidemann M, Putensen C, Popp J. Predisposing and precipitating factors of delirium after cardiac surgery: a prospective observational cohort study. Ann Surg. 2013 Jun;257(6):1160-7. doi: 10.1097/SLA.0b013e318281b01c. PMID 23426334
- [Result] Saczynski JS, Marcantonio ER, Quach L, Fong TG, Gross A, Inouye SK, Jones RN. Cognitive trajectories after postoperative delirium. N Engl J Med. 2012 Jul 5;367(1):30-9. doi: 10.1056/NEJMoa1112923. PMID 22762316
- [Result] Fong TG, Davis D, Growdon ME, Albuquerque A, Inouye SK. The interface between delirium and dementia in elderly adults. Lancet Neurol. 2015 Aug;14(8):823-832. doi: 10.1016/S1474-4422(15)00101-5. Epub 2015 Jun 29. PMID 26139023
- [Result] Turan A, Duncan A, Leung S, Karimi N, Fang J, Mao G, Hargrave J, Gillinov M, Trombetta C, Ayad S, Hassan M, Feider A, Howard-Quijano K, Ruetzler K, Sessler DI; DECADE Study Group. Dexmedetomidine for reduction of atrial fibrillation and delirium after cardiac surgery (DECADE): a randomised placebo-controlled trial. Lancet. 2020 Jul 18;396(10245):177-185. doi: 10.1016/S0140-6736(20)30631-0. PMID 32682483
- [Result] Angiulli F, Conti E, Zoia CP, Da Re F, Appollonio I, Ferrarese C, Tremolizzo L. Blood-Based Biomarkers of Neuroinflammation in Alzheimer's Disease: A Central Role for Periphery? Diagnostics (Basel). 2021 Aug 24;11(9):1525. doi: 10.3390/diagnostics11091525. PMID 34573867
- [Result] Grotti S, Falsini G. Delirium in cardiac patients. Eur Heart J. 2017 Aug 1;38(29):2244. doi: 10.1093/eurheartj/ehx380. No abstract available. PMID 28810719
- [Result] Muscat SM, Barrientos RM. The Perfect Cytokine Storm: How Peripheral Immune Challenges Impact Brain Plasticity & Memory Function in Aging. Brain Plast. 2021 Aug 23;7(1):47-60. doi: 10.3233/BPL-210127. eCollection 2021. PMID 34631420